CLINICAL TRIAL: NCT06451484
Title: Multicenter Study to Evaluate a Severity Score Using Venous MRI and CT in Patients With Post-Phlebitic Syndrome
Brief Title: Grade Analysis of Veins by MRI and CT in Post-Thrombotic Syndrome
Acronym: MR/CT PPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/04
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Lower Limb Venous Thrombosis
Keywords: post-thrombotic syndrome; CT; veins; MRI; severity score; multicenter study
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to improve the diagnosis of chronic lower limb venous thrombosis before a lower limb venous recanalization procedure. Additionally, if the MRI scores are comparable to those of the CT, MRI would reduce radiation exposure and limit the need for foot vein punctures that accompany CT use.

DETAILED DESCRIPTION:
Endovascular management of post-thrombotic syndrome (PTS) has created new opportunities for patients and interventional radiologists. PTS is the most chronic complication of deep vein thrombosis (DVT), occurring in 20% to 40% of patients despite optimal anticoagulant therapy within the first 1 to 2 years after a lower limb DVT. PTS is characterized by various symptoms lasting more than 6 months after a DVT, including mild pain or swelling, venous claudication, heaviness/fatigue, chronic pain or cramps, venous ulcers, edema, skin discoloration, and venous ectasia. Severe PTS negatively impacts quality of life. Several clinical tools or scales, such as the Villalta scale and CIVIQ-20, are used to diagnose and define PTS. Endovascular treatment of symptomatic chronic iliofemoral vein occlusions has shown good technical and clinical efficacy, with significant clinical benefits and improvements in the Villalta and CIVIQ scores. Proper planning of the recanalization procedure is essential, using CT and MRI imaging to analyze the venous anatomy in the pelvis, abdomen, and lower limbs. The CT is the reference examination for chronic lower limb thrombosis, performed using the Baldt technique to opacify the deep venous network and detect endoluminal adhesions. However, there are risks such as failure to puncture the veins on the back of the foot, pain during puncture, and flow artifacts. MRI is less commonly used due to its availability and long examination times, but its results are promising. The literature on chronic lower limb thrombosis is limited, with no consensus on lesion descriptions, highlighting the need for a descriptive lesion score

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged more than 18 years old,
* patient's oral consent,
* affiliated or beneficiary of health insurance

Exclusion Criteria:

* inability of the patient to understand the nature or risks or significance and implications of the clinical investigation,
* patient under legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had underwent MRI and/or phleboscan for chronic lower limb venous thrombosis
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Grade of vein severity on phleboscanner | Baseline
  Grade of vein severity on phleboscanner (from A-normal to D-very severe)

SECONDARY OUTCOMES:
Grade of vein severity on MRI | Baseline
  Grade of vein severity on MRI(from A-normal to D-very severe)
Inter-observator reproducibility on MRI | Baseline
  Intra-class correlation coefficient
Inter-observator reproducibility on phleboscan | Baseline
  Intra-class correlation coefficient
Reproducibility between MRI and phleboscan | Baseline
  Intra-class correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No